CLINICAL TRIAL: NCT02643576
Title: Designing a Food Benefit Program to Optimize Diet Quality for Obesity Prevention
Brief Title: Grocery Assistance Program Study
Acronym: GAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: DK098152; R01DK098152 (NIH)
Record Dates: First submitted 2014-12-22; First posted 2015-12-31 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Food Assistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): Usual SNAP-like food benefits
- Rewards (Experimental): Usual SNAP-like food benefits, plus a modification to this food benefit program that entails a 30% bonus on eligible fruit and vegetable purchases (i.e. F&V bonus)
  Interventions: Behavioral: F&V Bonus
- Restrictions (Experimental): Usual SNAP-like food benefits, plus a modification that requires no sugar-sweetened beverages, candy, or sweet baked goods be purchased
  Interventions: Behavioral: Restriction
- Rewards plus restrictions (Experimental): Usual SNAP-like food benefits, plus two modifications to this food benefit program: one modification includes a 30% bonus on eligible fruit and vegetable purchases and the other modification is that sugar-sweetened beverages, candy, or sweet baked goods are not allowed to be purchased (i.e. Bonus & Restriction)
  Interventions: Behavioral: Bonus & Restriction

INTERVENTIONS:
Behavioral: F&V Bonus — To examine the independent effect of offering an incentive (i.e. bonus dollars for fruit and vegetable purchases) to SNAP-like benefits to encourage the purchase of more healthful foods
  Arms: Rewards
Behavioral: Restriction — To examine the independent effect of prohibiting the use of SNAP-like benefits to purchase foods high in discretionary calories (i.e.sugar-sweetened beverages, candy, or sweet baked goods) on food purchases and diet quality
  Arms: Restrictions
Behavioral: Bonus & Restriction — To examine the joint effects of prohibiting the use of SNAP benefits to purchase foods high in discretionary calories and offering an incentive to encourage the purchase of more healthful foods
  Arms: Rewards plus restrictions

SUMMARY:
This highly innovative experimental trial is designed to examine the independent and joint effects of prohibiting the use of SNAP-like benefits to purchase foods high in discretionary calories and offering an incentive to encourage the purchase of more healthful foods.

DETAILED DESCRIPTION:
More than 1 in 10 Americans participate in the Supplemental Nutrition Assistance Program (SNAP), a Federal food and nutrition program administered by the United States Department of Agriculture (USDA). SNAP, formerly known as the Food Stamp Program, provides funds to low-income families for the purchase of food. Benefits are provided on an electronic benefits transfer (EBT) card that is used like an debit card at stores.

In recent years there has been growing recognition that SNAP participants are disproportionately obese, with poor diet contributing to this disparity. In response, there is great interest in considering ways in which SNAP may better meet its objective to help people and families buy the food they need for good health.

Modifications to SNAP currently under evaluation involve offering incentives to encourage participants to purchase more nutritious food items. There is concern, however, that this strategy alone may be of limited usefulness in improving the nutritional quality of the diet for obesity prevention because incentivizing the purchase of more nutritious foods does not necessarily reduce the purchase of less nutritious foods (substitution effect may not occur) and may even increase the total calories purchased.

An alternative strategy that has been extensively discussed by public health advocates and policy makers in recent years is prohibiting the purchase of less nutritious food items with SNAP benefits. Commonly consumed foods that are high in discretionary calories (defined as calories from solid fats, alcohol, and added sugars) are prime targets for exclusion because SNAP participants consume far more energy from discretionary calories (43%) than recommended. This strategy may be particularly effective if implemented in conjunction with incentives for the purchase of more nutritious foods.

No studies have been conducted to evaluate whether prohibiting the purchase of foods high in discretionary calories with SNAP benefits may improve diet quality and reduce risk of obesity. Likewise research is lacking on the effect of effect of pairing restrictions with incentives. Thus, we propose to pilot a highly innovative experimental trial designed to examine the independent and joint effects of prohibiting the use of SNAP benefits to purchase foods high in discretionary calories and offering an incentive to encourage the purchase of more healthful foods. Key indicators of feasibility will include recruitment and retention (are targeted number of participants recruited and retained at a high rate?); fidelity of the intervention (are compliance measures successfully collected and do they indicate close compliance with experimental condition assignment?); and completeness of baseline and follow-up data.

Using study data, analyses will be conducted to evaluate the independent and joint effects of prohibiting the use of SNAP benefits to purchase foods high in discretionary calories and offering an incentive to encourage the purchase of more nutritious foods.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Primary food shopper of household
* Not currently participating in the Supplemental Nutrition Assistance Program (SNAP)
* Not planning to apply for SNAP in the next 4 months
* Able to read and write in English
* ≤ 8 people living in household
* Have a gross monthly income level that places the household at or below 200 percent of the Federal poverty level for their household size.

Exclusion Criteria:

* < 18 years of age
* Not primary food shopper of household
* Currently participating in the Supplemental Nutrition Assistance Program (SNAP)
* Planning to apply for SNAP in the next 4 months
* Unable to read and write in English
* > 8 people living in household
* Have a gross monthly income level that places the household above 200 percent of the Federal poverty level for their household size

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Total Kilocalorie intake at 16 weeks | 16 weeks
  Evaluate the independent and joint effects on dietary intake of prohibiting the use of SNAP benefits to purchase foods high in discretionary calories and offering an incentive to encourage the purchase of more nutritious foods.
Change from baseline in reported levels of household food security at 16 weeks | 16 weeks
  Assessing any change from baseline in the score of the The U.S. Household Food Security Survey Module: Six-Item Short Form
Change from baseline in Healthy Eating Index (HEI) Score at 16 weeks | 16 weeks
  Evaluate the independent and joint effects on dietary intake of prohibiting the use of SNAP benefits to purchase foods high in discretionary calories and offering an incentive to encourage the purchase of more nutritious foods. More information about the HEI score can be found here: http://nccor.org/projects/hei/
Change from baseline in daily servings of fruits and vegetable (added together) at 16 weeks | 16 weeks
  Evaluate the independent and joint effects on dietary intake of prohibiting the use of SNAP benefits to purchase foods high in discretionary calories and offering an incentive to encourage the purchase of more nutritious foods.
  Servings of fruits and servings of vegetables are calculated from the output provided by NDS-R, which are based on the reported food intake as collected via 24-hour dietary recalls. Three recalls are collected at baseline and averaged; three recalls are collected at follow-up and averaged.
Change from baseline in daily total, in grams, of added sugars at 16 weeks | 16 weeks
  Evaluate the independent and joint effects on dietary intake of prohibiting the use of SNAP benefits to purchase foods high in discretionary calories and offering an incentive to encourage the purchase of more nutritious foods.

SECONDARY OUTCOMES:
Change from baseline in Body Mass Index | 16 weeks
  Evaluate the independent and joint effects on Body Mass Index of prohibiting the use of SNAP benefits to purchase foods high in discretionary calories and offering an incentive to encourage the purchase of more nutritious foods.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Harnack, DrPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota School of Public Health, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Valluri S, Mason SM, Peterson HH, French SA, Harnack LJ. The impact of financial incentives and restrictions on cyclical food expenditures among low-income households receiving nutrition assistance: a randomized controlled trial. Int J Behav Nutr Phys Act. 2021 Dec 4;18(1):157. doi: 10.1186/s12966-021-01223-7. PMID 34863192
- [Derived] French SA, Rydell SA, Mitchell NR, Michael Oakes J, Elbel B, Harnack L. Financial incentives and purchase restrictions in a food benefit program affect the types of foods and beverages purchased: results from a randomized trial. Int J Behav Nutr Phys Act. 2017 Sep 16;14(1):127. doi: 10.1186/s12966-017-0585-9. PMID 28915844
- [Derived] Harnack L, Oakes JM, Elbel B, Beatty T, Rydell S, French S. Effects of Subsidies and Prohibitions on Nutrition in a Food Benefit Program: A Randomized Clinical Trial. JAMA Intern Med. 2016 Nov 1;176(11):1610-1618. doi: 10.1001/jamainternmed.2016.5633. PMID 27653735
- See also: Brief Study Description & Study Contact Information — http://www.epi.umn.edu/gaps/